CLINICAL TRIAL: NCT04499859
Title: A Prospective, Multicenter, Randomized, Open-label Trial to Compare Low-dose ROSUvastatin Plus eZETimibe Versus High-dose Rosuvastatin in Patients With Acute Myocardial Infarction Undergoing Percutaneous Coronary Intervention
Brief Title: Low Dose Rosuvastatin Plus Ezetimibe Versus High-dose Rosuvastatin in AMI
Acronym: ROSUZET-AMI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kiyuk Chang, MD,PhD (Other)
Responsible Party: Sponsor-Investigator, Kiyuk Chang, MD,PhD, Professor of Medicine, The Catholic University of Korea
Organization: The Catholic University of Korea (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROSUZET-AMI
Record Dates: First submitted 2020-07-29; First posted 2020-08-05 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Myocardial Infarction; Statin Adverse Reaction; HMG-CoA Reductase Inhibitor Toxicity
MeSH Terms: conditions — Myocardial Infarction | interventions — Ezetimibe; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ezetimibe 10 mg plus rosuvastatin 5 mg (Experimental): Rosuzet 5/10 mg , once a day for 24 months
  Interventions: Drug: Ezetimibe 10mg + Rosuvastatin 5mg
- rosuvastatin 20 mg only (Active Comparator): Any brand drugs of rosuvastatin 20mg, once a day for 24 months
  Interventions: Drug: Rosuvastatin 20mg

INTERVENTIONS:
Drug: Ezetimibe 10mg + Rosuvastatin 5mg — Initial use of 10mg of ezetimibe combined with 5 mg of rosuvastatin
  Other Names: Rosuzet 10/5 mg
  Arms: ezetimibe 10 mg plus rosuvastatin 5 mg
Drug: Rosuvastatin 20mg — 20mg of Rosuvastatin as a standard treatment for AMI patients
  Other Names: Crestor 20mg
  Arms: rosuvastatin 20 mg only

SUMMARY:
Combination therapy of rosuvastatin 5mg and ezetimibe 10 mg showed similar achievement rate in decreasing LDL cholesterol level by 50% as single use of rosuvastatin 20 mg.

This trial aims to prove non-inferiority of concomitant usage of low dose rosuvastatin and ezetimibe among patients with acute myocardial infarction who went through percutaneous coronary intervention at decreasing major adverse cardiac events compared to the efficacy of single use of high dose rosuvastatin.

DETAILED DESCRIPTION:
IMPROVE-IT (Improved Reduction of Outcomes: Vytorin Efficacy International Trial) study showed that even when statin is not used as a treatment the rate of decrease of LDL cholesterol is correlated to the risk of heart disease. Yet whether concomitant use of ezetimibe and statin will have similar degree of clinical efficacy as single use of high dose statin in decreasing LDL cholesterol level needs further examination.

ELIGIBILITY:
Inclusion Criteria:

1. Adults Aged 19 and up
2. Patients diagnosed with myocardial infarction (both ST segment elevation and non-ST segment elevation) who were treated with percutaneous coronary intervention (Myocardial infarction defined as in the 4th Universal Definition of Myocardial Infarction)
3. For female patients who are of childbearing age, subjects that agreed on taking mandatory pregnancy test
4. Patients who agreed and signed on the informed consent form

Exclusion Criteria:

1. Patients with life expectancy of a year or less due to malignancy
2. Patients with chronic liver disease
3. Patients with sensitivity to active ingredient of the research drugs (ezetimibe and/or rosuvastatin) or patients who are prohibited to take ezetimibe and/or rosuvastatin.
4. Pregnant and/or breastfeeding
5. Female patients who are unable to use any means of contraception
6. Patients receiving hemodialysis, peritoneal dialysis patients and/or kidney transplant patients, due to end stage renal disease
7. Patients who participated in other clinical trial(s) within 3 months from the screening (except non-interventional observational study)
8. Patients considered inappropriate for the study for any other reason(s) by the inspector(s)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3548 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events (MACE) | 24 months
  A composite of cardiovascular death, major coronary events (non-fatal MI, documented unstable angina requiring hospital admission, all coronary revascularization with either PCI or bypass surgery occurring at least 30 days after randomization), or non-fatal stroke.

SECONDARY OUTCOMES:
death from any cause, a major coronary event, or a non-fatal stroke | 24 months
  death from any cause, a major coronary event, or a non-fatal stroke
cardiovascular death, non-fatal MI, or non-fatal stroke | 24 months
  cardiovascular death, non-fatal MI, or non-fatal stroke
all-cause death from any cause | 24months
cardiovascular death | 24months
any myocardial infaction | 24 months
any stroke | 24 months
any revascularization occurring at least 30 days after randomization | 24 months
LDL-C reduction <= 70mg/dl | 3 months
  LDL cholesterol level of 70mg/dL or less
LDL-C reduction <= 55mg/dl | 3 months
Rate of Statin associated muscle symptoms | 3 months
  Stain Associated Muscle Symptom questionnaire
drug discontinuation or dose reduction | 24 months
pill count drug adherence | 24 months
new onset diabetes | 24 months
cataract | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Kiyuk Chang, MD,PhD, Study Chair — Seoul St. Mary's Hospital
Locations (7):
- South Korea (7):
  - Bucheon St.Mary Hospital, Bucheon-si, Gyeonggido
  - St.Vincent's Hospital, Suwon, Gyeonggido
  - Uijeongbu St.Mary's Hospital, Uijeongbu-si, Gyeonggido
  - Daejeon St.Mary's Hospital, Daejeon
  - Incheon St.Mary's Hospital, Incheon
  - Seoul St.Mary's Hospital, Seoul
  - Yeouido St.Mary Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No
Aggregate summary data available on reasonable request. Exceptionally, and subject to Steering Committee approval, deidentified core analytic IPD may be accessed in a secure, non-downloadable virtual environment at the coordinating center. Contact PI (Kiyuk Chang) with proposal + ethics documentation; DUA required; costs may apply.

REFERENCES:
- [Derived] Choo EH, Kim CJ, Hwang BH, Lee KY, Oh GC, Lim S, Choi IJ, Kim DB, Kwon OS, Lee S, Choi Y, Park CS, Park MW, Kim HY, Lee HC, Kang TS, Sung JK, Woo SI, Park HS, Yun KH, Chang K; ROSUZET-AMI investigator. High-Intensity Statin versus Upfront Equivalent-Dose Combination of Moderate-Intensity Statin with Ezetimibe Following Acute Myocardial Infarction (ROSUZET-AMI): protocol of a multicentre, open-label, randomised non-inferiority trial. BMJ Open. 2025 Nov 5;15(11):e104127. doi: 10.1136/bmjopen-2025-104127. PMID 41198200